CLINICAL TRIAL: NCT04796389
Title: Result of a Music Intervention on Anxiety in Critically Ill Patients
Brief Title: Music for Anxiety in Critically Ill Patients
Acronym: RELACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Mathieu van der Jagt, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2020-0212
Record Dates: First submitted 2021-03-04; First posted 2021-03-12 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Anxiety
Keywords: music; anxiety; intensive care unit; critically ill
MeSH Terms: conditions — Anxiety Disorders; Critical Illness | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recorded music (Experimental): Recorded music intervention
  Interventions: Other: Music
- Control (No Intervention): Standard of care

INTERVENTIONS:
Other: Music — Preferred music of the participant administered using headphones.
  Arms: Recorded music

SUMMARY:
Rationale: Anxiety is common in critically ill patients, and has likely become more prevalent in the recent decade due to the imperative of the recent PADIS guidelines to use low levels of sedation and strive for wakefulness. Administration of sedative and analgesic medication is often chosen to reduce anxiety, especially when associated with agitation, but especially sedatives are associated with prolonged mechanical ventilation, delirium and muscle wasting and are therefore preferably minimized. Previous studies have suggested positive effects of music interventions on anxiety in the critically ill, next to other physiological signs such as pain. However, management of anxiety has not been included in the PADIS guidelines, and there is lack of evidence to treat it in spite of its growing importance. Therefore, we aim to study the effect of music intervention on anxiety in adult critically ill patients.

Objective: The primary objective is to assess the effect of music intervention on the level of anxiety.

Study design: A randomized controlled trial. Study population: Adult patients admitted to the intensive care unit, with whom communication is possible (Richmond Agitation Sedation Scale of -2 or higher).

Intervention (if applicable): The music group will be offered to listen to music two times per day for three days after inclusion, during 30-60 minutes per session. Chosen music will be based on the preference of the patient. The control group will receive standard of care during the entire study.

Main study parameters/endpoints: The primary outcome is the effect of music on the Visual Analogue Scale for anxiety (VAS-A). Secondary outcomes include effect of music on sedation and agitation level, medication requirement, pain, sleep, delirium, heart rate, mean arterial pressure, and ICU memory and experience.

ELIGIBILITY:
Inclusion Criteria:

* Patient is hemodynamically stable and communicable (RASS of -2 or higher in the 24h before intended inclusion: meaning patient is at least briefly awakened with eye contact to voice).
* Expected ICU stay upon randomisation of at least another 48 hours.
* Written informed consent acquired from the patient or legal representative.

Exclusion Criteria:

* Patients with severe hearing impairment, defined as no verbal communication possible.
* Neurological condition (e.g. severe stroke), when deemed to interfere with processing of music (e.g. not applicable to patients with minor stroke in past medical history without significant residual neurological deficits; those patients could be included).
* Insufficient knowledge of the Dutch or English language for informed consent.
* Participation in another study that may possibly intervene with the primary outcome measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Anxiety (VAS-A) | 1.5 year
  Measured using the Visual Analogue Scale for Anxiety (VAS-A), on a scale of 0 to 10, in which a higher score means a worse outcome.

SECONDARY OUTCOMES:
Anxiety (STAI-6) | 1.5 year
  Measured using the 6-item State- Trait Anxiety Inventory (STAI-6), on a scale of 20 to 80, in which a higher score means a worse outcome.
Sleep quality | 1.5 year
  Measured using a 7-item questionnaire, on a scale of 1 to 7, in which a lower score means a worse outcome.
Delirium | 1 year
  Measured with the Intensive Care Delirium Screening Checklist (ICDSC), on a scale of 0 to 8, in which a score of 4 or higher indicates delirium.
Sedative and opioid medication requirement | 1.5 year
  Including remifentanyl, propofol, benzodiazepines, dexmedetomidine, clonidine, paracetamol, sufentanyl, fentanyl, morphine, ketamine, epidural analgesia, haloperidol, and other benzodiazepines, atypical anxiolytics and antipsychotics.
ICU memory and experience | 1.5 year
  Assessed by the ICU memory tool (ICU-MT), difference is assessed per item.
Agitation and sedation level | 1.5 year
  Assessed using the Richmond- Agitation- Sedation Scale (RASS), on a scale of -5 to +4, negative scores indicate level of sedation (a more negative score indicates deeper sedation) and positive scores indicate levels of agitation (the higher the score the more agitated the patient).
Complications | 1.5 year
  Complications related to agitation, defined as removal of lines and tube by the patient.
Level of Pain | 1.5 year
  Measured using the Critical-Care Pain Observation (CPOT), on a scale of 0 to 8, in mechanically ventilated patients, or the NRS/VAS, on a scale of 0 to 10, for pain in non-ventilated and alert/oriented.
Heart Rate (HR) | 1.5 year
  Heart Rate at the time of anxiety assessment in beats per minute.
Mean Arterial Pressure (MAP) | 1.5 year
  Mean Arterial Pressure at the time of anxiety assessment in mmHg.

OTHER OUTCOMES:
ICU length of stay | 1.5 year
  Measured in total amount of hours spend in the ICU after inclusion.
Mechanical ventilation | 1.5 year
  Time spend on mechanical ventilation, measured in total amount of hours.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Dr. M. van der Jagt, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (3):
- Netherlands (3):
  - Erasmus MC, Rotterdam, South Holland
  - Ikazia, Rotterdam, South Holland
  - HagaZiekenhuis, The Hague, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kakar E, Ottens T, Stads S, Wesselius S, Gommers DAMPJ, Jeekel J, van der Jagt M. Effect of a music intervention on anxiety in adult critically ill patients: a multicenter randomized clinical trial. J Intensive Care. 2023 Aug 17;11(1):36. doi: 10.1186/s40560-023-00684-1. PMID 37592358
- [Derived] Kakar E, Van Mol M, Jeekel J, Gommers D, van der Jagt M. Study protocol for a multicentre randomised controlled trial studying the effect of a music intervention on anxiety in adult critically ill patients (The RELACS trial). BMJ Open. 2021 Oct 12;11(10):e051473. doi: 10.1136/bmjopen-2021-051473. PMID 34642197